A Single-arm Open-label Multicenter Clinical Study of Selinexor in Combination With HAD or CAG Rregimens in Relapsed or Refractory Acute Myeloid Leukemia

Project lead research unit: Shanxi Bethune Hospital

Version number: V2.0

Version date: 2022.11.3

**Board Status: Approved** 

Approval Number: YXLL-2022-134

Board Name: Ethics Committee of Shanxi Bethune

Hospital

Board Affiliation: Shanxi Bethune Hospital

#### Interventions:

#### 1. Treatment regimen:

Selinexor (60 mg) is used twice weekly for two weeks (four times, 240 mg total of selinexor) in combination with HAD or CAG regimens for reinduction therapy in patients with relapsed and refractory AML.

The two regimens combined with selinexor included:

(Bone marrow image indicates active hyperplasia) HAD regimen: homoharringtonine (HHT) (2mg/ m  $^2$ /d)×7days, daunorubicin (DNR, 40mg/ m  $^2$ /d)×3 days, cytarabine (Ara-C,100-200mg/ m  $^2$ /d)×7 days (no leukocyte-elevating drugs were applied throughout the course before and after treatment)

(Bone marrow image indicates hypoproliferation) CAG regimen: Granulocyte Colony-Stimulating Factor (G-CSF,  $5\mu g/kg/d$ , starting 12 hours before chemotherapy×14 days (d1-d14), aclacinomycin (20mg/d)×4 days (d1-4), cytarabine ( $10mg/m^2$ , subcutaneous injection, once every 12 hours)×14 days (d1-d14).

G-CSF was discontinued in the CAG regimen when WBC >20  $\times$  10 $^{9}$ /L, but chemotherapy was not stopped

### 2. Subsequent treatment regimen:

For patients eligible for allogeneic stem cell transplantation, stem cell transplantation is performed directly after treatment, and two courses (60 mg) of selinexor are maintained once a week and three weeks after transplantation;

Patients who are not eligible for transplantation or who have not undergone allogeneic stem cell transplantation should continue with two courses of treatment with HAD or CAG regimen, and selinexor (60 mg) is used once a week for two weeks.

# Supportive care:

- Platelet transfusion: Maintain platelet levels> 20 × 10<sup>9</sup>/L
- Red blood cell transfusion: keep hemoglobin> 80×10<sup>9</sup>/L
- Hepatoprotective drugs: routinely used in induction and consolidation therapy

## Bone marrow monitoring:

[Time point]: 10 times in total. These include bone puncture every 2 months at initial diagnosis, CR and consolidation maintenance period, and every 3 months after treatment until 2 years.

[Monitoring items]: monitoring of bone marrow morphology and molecular biology indicators.